CLINICAL TRIAL: NCT06431100
Title: Clinical Study on the Safety and Efficacy of GK01 Autologous Tumor-reactive T Cells (TRT) in Patients With Advanced Solid Tumors
Brief Title: a Single-arm, Single-center, Open Clinical Study
Acronym: GK-01
Status: Recruiting | Type: Observational
Sponsor: Beijing Geekgene Technology Co., LTD (Industry)
Responsible Party: Sponsor
Other Study IDs: GK-01
Record Dates: First submitted 2024-05-20; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Gastric Cancer; Esophageal Cancer; Cervical Cancer; Non-Small Cell Lung Cancer NSCLC; Triple Negative Breast Cancer TNBC
Keywords: TRT; cell therapy; advanced tumor; safety; efficiency; adverse event
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cell therapy interventional single arm: According to the cell transfusion protocol, GK01 cells were given at a certain dose level to observe the safety and tolerability of the patients after the transfusion, explore the pharmacokinetic/pharmacodynamic characteristics after the transfusion, and preliminarily evaluate the effectiveness of the experimental drug GK01 cells according to the RECIST 1.1 standard.
  Interventions: Biological: TCR T-cells

INTERVENTIONS:
Biological: TCR T-cells — The strengthened T cells are re-infused into the patient to achieve the killing effect

SUMMARY:
This trial plans to enroll many patients with advanced solid tumors to complete GK01 cell transfusion, including but not limited to advanced gastric cancer, esophageal cancer, cervical cancer, triple-negative breast cancer, and non-small cell lung cancer. For patients with advanced solid tumors eligible for inclusion, autologous tumor-reactive T cells (experimental drug GK01) were cultured and prepared, and a certain dose of GK01 cells was given according to the cell transfusion plan, and the safety and tolerability of the patients after transfusion were observed. Exploratory evaluation of pharmacokinetic/pharmacodynamic profiles following reinfusion and initial evaluation of efficacy of investigational drug GK01 cells according to RECIST 1.1 criteria.

ELIGIBILITY:
Inclusion Criteria:

* Participants who meet all of the following criteria are eligible for admission to the study:

  1. 18≤ age ≤75 years old, male or female;
  2. Patients with incurable advanced gastric cancer, esophageal cancer, cervical cancer, triple-negative breast cancer, non-small cell lung cancer, and other malignancies who have failed standard treatment (standard treatment failure is defined as those treated according to the 2022 CSCO Guidelines and whose tumor efficacy is assessed as disease progression (PD) or tumor recurrence or inability to tolerate existing treatment options);
  3. There are tumor tissues or cancerous exudative thoracoabdominal fluid that can be used to isolate TRTs: the total volume of the solid tissue taken must be > 0.5cm3 or the weight must be >0.5g, the cancerous exudative thoracoabdominal fluid taken should contain at least 5×10^8 total cells, and the lesions taken have not been treated with oncolytic virus.
  4. There is at least one measurable lesion (according to RECIST1.1 criteria) even after TRTs sampling/puncture biopsy;
  5. ECOG score 0-1;
  6. The expected survival period is greater than 3 months;
  7. Sufficient hematology and end-organ function, as defined by the following laboratory test results, should be completed within 14 days prior to TRTs tumor tissue collection:

     1. Blood routine: white blood cell count ≥2.5×10^9/L; Absolute neutrophil count (ANC) ≥1.5×10^9/L; Absolute lymphocyte count (ALC) ≥1.0×10^9/L; Platelet (PLT) ≥80×10^9/L; Hemoglobin (HGB) ≥90g/L;
     2. Coagulation function: International standardized ratio of prothrombin time (INR) ≤1.5×ULN; Partial prothrombin time (APTT) ≤1.5×ULN, unless anticoagulant therapy has been received within the previous 7 days;
     3. Renal function: serum creatinine ≤1.5mg/dL (or 132.6μmol/L) or creatinine clearance ≥60mL/ min;
     4. Liver function: aspartate aminotransferase (AST/SGOT) ≤3×ULN; Alanine transaminase (ALT/SGPT) ≤3×ULN; Total bilirubin (TBIL) ≤1.5×ULN; Note: In patients with liver metastasis or primary liver tumor, aspartate and alanine aminotransferase should be ≤5×ULN; For patients with a history of Gilbert syndrome or suspected Gilbert syndrome, total bilirubin (TBIL) should be ≤3×ULN;
     5. Urine routine: urinary protein <2+, or 24-hour urinary protein quantity <1g;
     6. Left ventricular ejection fraction (LVEF) ≥50% by echocardiography;
     7. Pulmonary function tests with FEV1>60% or FEV1/FVC>0.7;
     8. Blood oxygen saturation ≥ 93%.
  8. Women of childbearing age who have a negative urine pregnancy test during screening and baseline and agree to use highly effective contraception for at least 1 year after the infusion; Male subjects whose partners are fertile must agree to use effective contraceptive methods and refrain from sperm donation for at least 1 year after the infusion;
  9. No absolute or relative contraindications to surgery or puncture;
  10. Any treatment for malignant tumors, including radiotherapy, chemotherapy, endocrine therapy, targeted therapy, tumor embolization, or Chinese medicine/herbal therapy with anti-tumor indications, must be discontinued 7 days before TRT sampling;
  11. Sign a written informed consent (ICF) voluntarily, and have good compliance with the protocol requirements for visits or planned visits and other relevant research procedures.

Exclusion Criteria:

* Subjects who meet any of the following criteria will not be eligible to participate in this clinical trial:

  1. Prior allergy to cyclophosphamide, fludarabine and interleukin-2 contraindications or to any component of the infusion product formulation or to other drugs to be used during the study (antibiotics, human serum albumin, dextran 40, etc.);
  2. Any NCI CTCAE5.0 immune-related adverse reaction (irAE) grade >3 that has been permanently discontinued during any previous immunotherapy;
  3. Patients with prior primary immunodeficiency and active autoimmune disease;
  4. Previous history of organ allotransplantation, allogeneic stem cell transplantation and kidney replacement therapy;
  5. Patients with current or past irreversible interstitial lung disease (except those caused by radiotherapy);
  6. Combined with 2 or more malignant tumors; (Except for the following cases: malignant tumors that have been cured, such as non-melanoma skin cancer and in situ cervical cancer, bladder cancer, breast cancer, thyroid cancer, etc. that have survived more than 5 years without disease.)
  7. Uncontrolled co-morbidity includes, but is not limited to, uncontrolled hypertension (systolic blood pressure ≥160mmHg and/or diastolic blood pressure ≥100mmHg) even after standard treatment, or any unstable cardiovascular and cerebrovascular disease, including transient ischemic attack, cerebrovascular accident, myocardial infarction, and unstable angina pectoral, that has occurred in the 6 months prior to treatment induction; Congestive heart failure rated III or IV by the New York Heart Association (NYHA); Ejection fraction < 50%; Severe heart rhythm or conduction abnormalities, such as ventricular arrhythmias requiring clinical intervention, degree II-III atrioventricular block, etc. Electrocardiogram results show clinically significant abnormalities, or QTcF≥450ms (if the first examination is abnormal, the interval of at least 5 minutes, retest twice, using the comprehensive result/average value to judge eligibility);
  8. Patients with esophageal or gastric varices that require immediate intervention (such as ligation or sclerotherapy) or are considered by the investigator or gastroenterologist or hepatologist to be at high risk of bleeding, have evidence of portal hypertension (including splenomegalysis on imaging), or have a history of varicose bleeding must undergo endoscopic evaluation within 3 months prior to enrollment;
  9. Uncontrolled metabolic disorders, such as in patients with diabetes, or other non-malignant organ or systemic disease or cancer secondary reactions that can lead to higher medical risk and/or uncertainty in the evaluation of survival;
  10. Hepatic encephalopathy, hepatorenal syndrome or Child-Pugh grade C or more severe cirrhosis, liver failure;
  11. Clinically uncontrollable third space effusion, such as pleural fluid and ascites that could not be controlled by drainage or other methods before enrollment;
  12. Combined with other serious organic disease or mental illness;
  13. Patients with central nervous system metastasis;
  14. Uncontrolled systemic active infection;
  15. Receive vaccination within 2 months before signing the informed consent, or plan to receive vaccination during the study;
  16. Currently or within 30 days before signing the informed consent to participate in clinical trials of other drugs or biotherapeutics, except cell therapy that has been fully metabolized;
  17. have used within 4 weeks prior to the treatment, or have concomitant disease or active autoimmune disease that the investigator determined required the use of glucocorticoids or other immunosuppressive drugs during the trial period, excluding local percutaneous absorption of glucocorticoids (i.e., no more than 5 mg/ day of prednisone or equivalent doses of other glucocorticoids);
  18. Surgical treatment, interventional therapy, radiotherapy, chemotherapy and immunotherapy for the studied disease were performed within 2 weeks before the treatment;
  19. HIV positive, serological test positive for syphilis, or clinically active hepatitis B or C, including carriers of the virus (for hepatitis B, HBsAg positive persons should be excluded; For hepatitis C, HCVAB-positive patients need to be excluded);
  20. Women who are breastfeeding during pregnancy or lactation;
  21. Poor compliance due to physiological, family, social, geographical and other factors, unable to cooperate with the study protocol and follow-up plan;
  22. Other conditions deemed unsuitable for participation in this experiment by the researcher.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: GK01 cell transfusions were performed in 10 patients with advanced solid tumors, including but not limited to advanced non-small cell lung cancer, gastric cancer, and esophageal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-07-19 (Actual); Primary Completion 2026-07-19 (Estimated); Study Completion 2026-11-19 (Estimated)

PRIMARY OUTCOMES:
safety and tolerability | From enrollment to the end of follow-up visit at 22weaks or more
  To evaluate the safety and tolerability of GK01 autologous tumor-reactive T cells (TRT) in patients with advanced solid tumors.

SECONDARY OUTCOMES:
specificity and persistence | From enrollment to the end of treatment at 28 days
  To explore the specificity and persistence of GK01 autologous tumor-reactive T cells (TRT) expansion in patients with advanced solid tumors
initial efficacy | From enrollment to the end of treatment at 28 days
  To evaluate the initial efficacy of GK01 autologous tumor-reactive T cells (TRT) in the treatment of patients with advanced solid tumors based on RECIST 1.1 criteria

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided